CLINICAL TRIAL: NCT00246376
Title: Diet/Exercise, Niacin, Fenofibrate for HIV Lipodystrophy
Brief Title: Diet, Exercise, Niacin, and Fenofibrate to Reduce Heart Disease Risk Factors in Individuals With HIV Lipodystrophy or Dyslipidemia
Acronym: HeartPositive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Legacy Community Health Center (Unknown)
Responsible Party: Principal Investigator, Ashok Balasubramanyam, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-14105; R01HL073696 (NIH)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; HIV Infections; Hyperlipidemia; Hypertriglyceridemia; Insulin Resistance; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; HIV Infections; Hyperlipidemias; Hypertriglyceridemia; Insulin Resistance; Atherosclerosis | interventions — Diet; Exercise; Niacin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Placebo Comparator): Subjects receive lifestyle advice and placebos for Niaspan and Tricor
  Interventions: Other: Placebos
- 2 (Experimental): Diet, exercise, and two placebos
  Interventions: Behavioral: Diet; Behavioral: Exercise; Other: Placebos
- 3 (Experimental): Diet, exercise, Niaspan, and placebo
  Interventions: Behavioral: Diet; Behavioral: Exercise; Drug: Niacin; Other: Placebos
- 4 (Experimental): Diet, exercise, placebo, and Tricor
  Interventions: Behavioral: Diet; Behavioral: Exercise; Drug: Fenofibrate; Other: Placebos
- 5 (Experimental): Diet, exercise, Niaspan, and Tricor
  Interventions: Behavioral: Diet; Behavioral: Exercise; Drug: Niacin; Drug: Fenofibrate

INTERVENTIONS:
Behavioral: Diet — ATP-III diet
  Arms: 2; 3; 4; 5
Behavioral: Exercise — Supervised exercise in study gym
  Arms: 2; 3; 4; 5
Drug: Niacin — Niaspan, titrated up to 2 grams per day
  Arms: 3; 5
Drug: Fenofibrate — Tricor, 120 mg per day
  Arms: 4; 5
Other: Placebos — Placebos for Niaspan and Tricor
  Arms: 1; 2; 3; 4

SUMMARY:
This study will evaluate the efficacy of diet and exercise (DE), with and without niacin and fenofibrate, in reducing the cardiovascular risk of patients with HIV lipodystrophy or dyslipidemia.

DETAILED DESCRIPTION:
BACKGROUND:

HIV lipodystrophy syndrome is associated with both metabolic (e.g., dyslipidemia and insulin resistance) and anthropomorphic (e.g., lipoatrophy and central obesity) abnormalities. These defects are likely to predispose HIV patients on highly active antiretroviral therapy (HAART) to accelerated cardiovascular morbidity. Based on studies of key mechanisms of altered lipid kinetics in these patients, evidence that DE patterns of patients with HIV lipodystrophy are inadequate to manage cardiovascular risk factors, and current recommendations for treatment of atherosclerosis and insulin resistance, the following is hypothesized: 1) an intensive lifestyle intervention with DE will improve the plasma lipid profile, decrease visceral fat mass, and improve hormonal, metabolic, and lipoprotein markers associated with insulin resistance; and 2) adding niacin, fenofibrate, or a combination of the two drugs to the intensive lifestyle intervention will result in further improvement in the cardiovascular risk profile.

DESIGN NARRATIVE:

This randomized, placebo-controlled study of 200 hypertriglyceridemic HIV patients on stable HAART treatment has the following specific aims: 1) to compare the effects of usual care, intensive DE, DE plus niacin, DE plus fenofibrate, and DE plus niacin plus fenofibrate on fasting plasma lipid concentrations (primary endpoint); 2) to compare the effects of the five treatment protocols on body fat distribution; and 3) to compare the effects of the five treatment protocols on hormonal, lipoprotein, and metabolic markers of insulin resistance. The collaborative team has expertise in lipid and lipoprotein metabolism, innovative and effective diet modification programs, intensive exercise programs in HIV patients, and studies of antilipidemic and antiretroviral agents. Therefore, this study will determine the efficacy of DE, with and without niacin and fenofibrate, in reducing the cardiovascular risk of patients with HIV lipodystrophy or dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* On stable HAART regimen for at least 6 months prior to study entry
* T-cell count greater than 100 and viral load less than 1,000 for at least 6 months prior to study entry
* Fasting triglyceride level greater than 150 mg/dl
* Body mass index (BMI) greater than 18.5 and less than 30
* Uses barrier contraception

Exclusion Criteria:

* Fasting triglyceride level greater than 1000 mg/dl
* BMI less than 18.5 or greater than 30
* Taking diabetic medication or HbA1c less than 7.0
* Use of lipid lowering medication in the 30 days prior to study entry
* Unable to exercise
* T-cell count less than 100
* Current medical condition that makes exercise unadvisable
* History of coronary artery disease (CAD)
* Use of dietary supplements (within 30 days of study entry) that may affect lipid levels including, but not limited to, the following:

  1. Omega-3 fatty acids
  2. L-Carnitine
  3. Soluble fiber supplements
  4. Guggul
  5. Garlic supplements
  6. Niacin greater than 25mg/d
  7. Oral liquid supplements
* Use of steroids, hormones, or testosterone (without diagnosis of hypogonadism, testosterone less than 300 ng/dl)
* Irregular periods
* Depo-Provera
* Hypo- or Hyperthyroidism
* Adrenal insufficiency
* Serum alanine or aspartate aminotransferase level greater than 3 times the upper limit of normal
* Alcohol abuse
* Renal insufficiency (creatinine level greater than 1.5 mg/dl)
* Coumadin therapy
* Pregnancy
* Peptic ulcer disease
* Cholelithiasis
* History of hyperuricemia
* History of myositis or rhabdomyolysis
* Known adverse reaction to niacin or fibrates
* Hepatitis C therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2004-01; Primary Completion 2009-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Balasubramanyam, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Samson SL, Pownall HJ, Scott LW, Ballantyne CM, Smith EO, Sekhar RV, Balasubramanyam A. Heart positive: design of a randomized controlled clinical trial of intensive lifestyle intervention, niacin and fenofibrate for HIV lipodystrophy/dyslipidemia. Contemp Clin Trials. 2006 Dec;27(6):518-30. doi: 10.1016/j.cct.2006.07.002. Epub 2006 Jul 21. PMID 16914390
- [Result] Balasubramanyam A, Coraza I, Smith EO, Scott LW, Patel P, Iyer D, Taylor AA, Giordano TP, Sekhar RV, Clark P, Cuevas-Sanchez E, Kamble S, Ballantyne CM, Pownall HJ. Combination of niacin and fenofibrate with lifestyle changes improves dyslipidemia and hypoadiponectinemia in HIV patients on antiretroviral therapy: results of "heart positive," a randomized, controlled trial. J Clin Endocrinol Metab. 2011 Jul;96(7):2236-47. doi: 10.1210/jc.2010-3067. Epub 2011 May 11. PMID 21565796
- [Derived] Gillard BK, Raya JL, Ruiz-Esponda R, Iyer D, Coraza I, Balasubramanyam A, Pownall HJ. Impaired lipoprotein processing in HIV patients on antiretroviral therapy: aberrant high-density lipoprotein lipids, stability, and function. Arterioscler Thromb Vasc Biol. 2013 Jul;33(7):1714-21. doi: 10.1161/ATVBAHA.113.301538. Epub 2013 May 2. PMID 23640486
- [Derived] Vu CN, Ruiz-Esponda R, Yang E, Chang E, Gillard B, Pownall HJ, Hoogeveen RC, Coraza I, Balasubramanyam A. Altered relationship of plasma triglycerides to HDL cholesterol in patients with HIV/HAART-associated dyslipidemia: further evidence for a unique form of metabolic syndrome in HIV patients. Metabolism. 2013 Jul;62(7):1014-20. doi: 10.1016/j.metabol.2013.01.020. Epub 2013 Mar 19. PMID 23522788
- [Derived] Wooten JS, Nambi P, Gillard BK, Pownall HJ, Coraza I, Scott LW, Nambi V, Ballantyne CM, Balasubramanyam A. Intensive lifestyle modification reduces Lp-PLA2 in dyslipidemic HIV/HAART patients. Med Sci Sports Exerc. 2013 Jun;45(6):1043-50. doi: 10.1249/MSS.0b013e3182843961. PMID 23299761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited mainly from the Legacy Community Health Center and Thomas Street Clinic of the Harris County Hospital District and from Houston Area Community Services and private clinics. Recruitment period: January 2004 to September 2009.
Pre-assignment Details: If potential subjects were taking nutritional supplements or lipid-lowering drugs, these were discontinued for washout for 6 weeks - baseline fasting lipid levels were then measured to determine eligibility prior to randomization.
Groups:
- Group 1: Usual Care: Subjects receive lifestyle advice and placebos for Niaspan and Tricor
- Group 2: Diet / Exercise: Diet, exercise, and two placebos
- Group 3: Diet / Exercise + Fenofibrate: Diet, exercise, Fenofibrate, and Niaspan placebo
- Group 4: Diet / Exercise + Niacin: Diet, exercise, Fenofibrate placebo, and Niaspan
- Group 5: Diet / Exercise + Niacin + Fenofibrate: Diet, exercise, Fenofibrate and Niaspan
Period: Overall Study
Arm/Group | Group 1: Usual Care | Group 2: Diet / Exercise | Group 3: Diet / Exercise + Fenofibrate | Group 4: Diet / Exercise + Niacin | Group 5: Diet / Exercise + Niacin + Fenofibrate
Started | 41 | 43 | 45 | 47 | 45
After Dietary run-in at Two Weeks | 30 | 38 | 41 | 40 | 42
Completed | 26 | 24 | 29 | 21 | 28
Not Completed | 15 | 19 | 16 | 26 | 17
Not completed — Dropped/withdrew during dietary run-in | 11 | 5 | 4 | 7 | 3
Not completed — Adverse Event | 2 | 3 | 1 | 3 | 1
Not completed — Lost to Follow-up | 2 | 11 | 11 | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Usual Care | Group 2: Diet / Exercise | Group 3: Diet / Exercise + Fenofibrate | Group 4: Diet / Exercise + Niacin | Group 5: Diet / Exercise + Niacin + Fenofibrate | Total
Number analyzed (Participants) | 41 | 43 | 45 | 47 | 45 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 43 | 45 | 47 | 45 | 220
  >=65 years | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 9 | 5 | 7 | 29
  Male | 37 | 39 | 36 | 42 | 38 | 192
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 45 | 47 | 45 | 221

OUTCOME MEASURES:

1. Primary Outcome: Triglycerides
Description: Triglycerides (mg/dL): Fasting lipid levels
Time Frame: Measured at 24 weeks
Population: All those who underwent the 2-week (first follow-up) measurement and continued in the study.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Group 1 - Usual Care: These subjects did not participate in the diet/exercise program and took placebos.
- Group 2 - Diet/Exercise Only: These subjects participated in the diet/exercise program and took placebos.
- Group 3 - Diet/Exercise + Fenofibrate: These subjects participated in the diet/exercise program and took active fenofibrate + niacin placebo.
- Group 4 - Diet/Exercise + Niacin: These subjects participated in the diet/exercise program and took active niacin + fenofibrate placebo.
- Group 5 - Diet/Exercise + Fenofibrate + Niacin: These subjects participated in the diet/exercise program and took active fenofibrate + active niacin.
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 30 | 38 | 41 | 40 | 42
mg/dL | 199 (24.9) | 216.9 (28.6) | 155.1 (18.5) | 177.6 (24.2) | 135.6 (16.9)

2. Secondary Outcome: Insulin Sensitivity
Description: Adiponectin (micrograms/ml)
Time Frame: Measured at 24 weeks
Population: All subjects who completed 24 weeks.
Measure: Mean (Standard Error); unit: micrograms/ml
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 26 | 24 | 29 | 21 | 28
micrograms/ml
  Fasting insulin | 8.7 (2) | 6.7 (1.6) | 9.5 (1.6) | 11.9 (3) | 10.3 (2.5)
  HOMA-IR | 1.92 (0.47) | 1.38 (0.36) | 2.02 (0.47) | 2.76 (0.75) | 2.38 (0.62)
  Insulin sensitvity index | 3.54 (0.73) | 4.95 (1.1) | 3.81 (0.76) | 2.88 (0.67) | 2.38 (0.62)
  Adiponectin | 7.12 (1.09) | 6.04 (0.98) | 5.24 (0.76) | 11.01 (1.87) | 10.34 (1.67)

3. Secondary Outcome: Body Composition
Description: 1. Body cell mass (kg)
  2. Fat mass (kg)
Time Frame: Measured at 24 weeks
Population: The number corresponds to the number of subjects who completed the study (see Participant flow)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 26 | 24 | 29 | 21 | 28
kg
  Body cell mass | 59.6 (2.3) | 67.3 (2) | 66.6 (1.8) | 67.1 (2.1) | 68.2 (2)
  Fat mass | 36.8 (1.9) | 37.5 (1.6) | 35.8 (1.5) | 37.7 (1.8) | 36.2 (1.7)

4. Primary Outcome: Non-HDL-C
Description: non-HDL-C (mg/dL): Fasting lipid levels
Time Frame: Measured at 24 weeks
Population: All those who underwent the 2-week (first follow-up) measurement and continued in the study.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 30 | 38 | 41 | 40 | 42
mg/dl | 162.2 (7.8) | 165.4 (8.1) | 145.8 (7.4) | 154 (8.3) | 137.1 (7.7)

5. Primary Outcome: HDL-C
Description: HDL-C (mg/dL): Fasting lipid levels
Time Frame: Measured at 24 weeks
Population: All those who underwent the 2-week (first follow-up) measurement and continued in the study.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 30 | 38 | 41 | 40 | 42
mg/dl | 37.1 (1.8) | 38.7 (1.9) | 40.7 (1.8) | 41.8 (2.2) | 44.8 (2.1)

6. Primary Outcome: Total Cholesterol
Description: Total cholesterol (mg/dL): Fasting lipid levels
Time Frame: Measured at 24 weeks
Population: All those who underwent the 2-week (first follow-up) measurement and continued in the study.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 30 | 38 | 41 | 40 | 42
mg/dL | 195.6 (7.7) | 200.1 (8.3) | 184 (6.9) | 190.8 (8.2) | 178.4 (7)

7. Primary Outcome: Total Cholesterol : HDL-C Ratio
Description: Total cholesterol : HDL-C ratio: Fasting lipid levels
Time Frame: Measured at 24 weeks
Population: All those who underwent the 2-week (first follow-up) measurement and continued in the study.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Group 1 - Usual Care | Group 2 - Diet/Exercise Only | Group 3 - Diet/Exercise + Fenofibrate | Group 4 - Diet/Exercise + Niacin | Group 5 - Diet/Exercise + Fenofibrate + Niacin
Number analyzed (Participants) | 30 | 38 | 41 | 40 | 42
ratio | 5.2 (0.3) | 5.1 (0.3) | 4.5 (0.2) | 4.6 (0.3) | 4 (0.2)

ADVERSE EVENTS:
Time Frame: Throughout duration of study (5 years)
Arm/Group | Group 1: Usual Care | Group 2: Diet / Exercise | Group 3: Diet / Exercise + Fenofibrate | Group 4: Diet / Exercise + Niacin | Group 5: Diet / Exercise + Niacin + Fenofibrate
Serious Adverse Events (participants affected / at risk) | 7/30 | 10/38 | 6/41 | 4/40 | 5/42
Other Adverse Events (participants affected / at risk) | 17/30 | 11/38 | 12/41 | 33/40 | 25/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Usual Care (N=30) | Group 2: Diet / Exercise (N=38) | Group 3: Diet / Exercise + Fenofibrate (N=41) | Group 4: Diet / Exercise + Niacin (N=40) | Group 5: Diet / Exercise + Niacin + Fenofibrate (N=42)
Transaminases elevated >3 times upper normal limit (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Chest pain / angina (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Serum creatining > 1.5 mg/dL (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Triglycerides > 1000mg/dl (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) — hypertriglyceridemia
Elevated Bilirubin (Hepatobiliary disorders) | 3 (3) | 5 (5) | 4 (4) | 0 (0) | 2 (2) — Elevated Bilirubin
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Usual Care (N=30) | Group 2: Diet / Exercise (N=38) | Group 3: Diet / Exercise + Fenofibrate (N=41) | Group 4: Diet / Exercise + Niacin (N=40) | Group 5: Diet / Exercise + Niacin + Fenofibrate (N=42)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash/Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 16 (16) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Body ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Loss of appetite (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
High dropout rate, especially by loss to follow-up (with no explanation). Flushing was common among patients taking niacin, and this (with transportation and socio-economc problems) could have contributed to the high drop-out rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No